CLINICAL TRIAL: NCT01843946
Title: Clinical Efficacy of Roxithromycin in Men With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Hyun-Sop Choe, Doctor, The Catholic University of Korea
Other Study IDs: Rulid-2011
Record Dates: First submitted 2013-04-27; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Prostatitis; Chronic Pelvic Pain Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Roxithromycin is effective in the treatment of intracellular organisms, including chlamydia and mycoplasma, and exhibits anti-inflammatory and immunomodulatory effects on respiratory diseases. To explore the potential therapeutic benefit of roxithromycin in chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS), this study compared the effect of roxithromycin with ciprofloxacin and aceclofenac.

DETAILED DESCRIPTION:
A total of 75 patients with CP/CPPS were randomized to three groups in open-label: group 1, ciprofloxacin; group 2, aceclofenac; and group 3, roxithromycin. The patients were treated for 4 weeks and were subsequently followed for 12 weeks. Changes from baseline in the total and domain scores of the NIH Chronic Prostatitis Symptom Index (NIH-CPSI) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of category IIIa of IIIb chronic prostatitis
* NIH-CPSI (National Institute of Health Chronic Prostatitis Symptom Index) score ≥ 15

Exclusion Criteria:

* Urinary tract infection or uropathogen within the past 12 months
* Serious medical problems
* NIH consensus exclusion criteria13 (presence of active urethritis, urogenital cancer, urinary tract disease, functionally significant urethral stricture, neurological disease affecting the bladder, etc.)
* Drug therapy that might affect lower urinary tract functions within the past 3 months

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 75
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
NIH-CPSI score | 12 weeks
  Changes from baseline in the total and domain scores of the NIH Chronic Prostatitis Symptom Index (NIH-CPSI) were evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Sop Choe, Dr, Principal Investigator — Saint Vincent's Hospital, Korea
Locations (1):
- The Catholic University of Korea, St. Vincent's Hospital, Suwon, South Korea

REFERENCES:
- [Derived] Choe HS, Lee SJ, Han CH, Shim BS, Cho YH. Clinical efficacy of roxithromycin in men with chronic prostatitis/chronic pelvic pain syndrome in comparison with ciprofloxacin and aceclofenac: a prospective, randomized, multicenter pilot trial. J Infect Chemother. 2014 Jan;20(1):20-5. doi: 10.1016/j.jiac.2013.07.010. Epub 2013 Dec 11. PMID 24462419